CLINICAL TRIAL: NCT06380270
Title: Study to Evaluate the Safety and Human Tolerance of the Oral Probiotic Streptococcus Salivarius eK12: A Randomized, Double-blind Clinical Trial
Brief Title: Evaluation of Safety and Human Tolerance of Oral Probiotic Streptococcus Salivarius eK12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MMC/ERC/03.03.2025
Record Dates: First submitted 2024-04-14; First posted 2024-04-23 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Safety; Tolerability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic supplement group (Experimental): Participants in this arm will daily receive 2 orally dissolving tablets (single administration) of probiotic Streptococcus salivarius eK12 (Bactoblis® EVOL: containing ca. 10 billion CFU of S. salivarius eK12) for 28-days.
  Interventions: Dietary Supplement: Oral probiotic Streptococcus salivarius eK12
- Control group (Placebo Comparator): Participants in this arm will daily receive 2 orally dissolving placebo tablets (single administration) for 28-days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Oral probiotic Streptococcus salivarius eK12 — Bactoblis® EVOL (containing 10 billion CFU of S. salivarius eK12)
  Arms: Probiotic supplement group
Other: Placebo — Orally dissolving placebo tablets
  Arms: Control group

SUMMARY:
The human oral cavity contains a diverse community of microorganisms essential for oral and overall health. Streptococcus salivarius K12 (eK12) has emerged as a promising oral probiotic due to its natural colonization of the throat and its ability to inhibit pathogens such as Streptococcus pyogenes, a major cause of streptococcal pharyngitis. It supports oral hygiene by producing antimicrobial substances like salivaricins and inhibiting odor-causing bacteria. The engineered eK12 variant (Bactoblis® Evol) has been developed to overcome inactivation by GAS-secreted protease SpeB, thereby enhancing its prophylactic potential against Group A Streptococcus (GAS) colonization.

This clinical study includes a randomized, double-blind, placebo-controlled trial in Pakistan to evaluate the safety and human tolerance of eK12 in healthy adults. To enhance generalizability, an additional open-label cohort of healthy adults in Italy will receive eK12 without a control group.

DETAILED DESCRIPTION:
The aim of the present clinical study is to evaluate the safety and tolerability of Streptococcus salivarius eK12 in healthy adults. The study consists of a randomized, double-blind, placebo-controlled arm in Pakistan involving 29 participants (allocated 1:1 to eK12 or placebo).

In addition, an open-label cohort of 20 healthy adults will be enrolled in Italy, all of whom will receive eK12, to assess tolerability in a separate population without a control group. This complementary cohort is included to enhance the generalizability of the findings across different populations and to obtain supportive safety data in a real-world setting where the product (commercially available in the EU as Bactoblis® Evol) is already in use.

Through comprehensive assessments and close monitoring of participants, this study will provide critical insights into the safety profile and human tolerance of the probiotic-modified strain. The findings will contribute to the growing body of knowledge needed to support its use in oral health management.

ELIGIBILITY:
Inclusion Criteria:

* Adults, both male and female, aged 18 to 60 years.
* Stable health condition with no acute illness at the time of enrollment.
* BMI 18.5-35 kg/m2
* No known food allergies or intolerances to probiotics
* All clinical chemistry, hematology and urinalysis parameters and vital signs (blood pressure, respiratory rate, temperature, heart rate) within clinically acceptable ranges.
* Ability and willingness to provide informed consent.
* Must be willing to comply with study procedures and attend scheduled visits.

Exclusion Criteria:

* Individuals with a history of severe allergies or adverse reactions to probiotics or any of the components of the study product.
* Participants with a recent history of oral surgery or dental procedures within the past 4 weeks.
* Individuals with severe dental problems or undergoing active dental treatment.
* Individuals with a known diagnosis of systemic diseases affecting the oral cavity (e.g., oral cancer, Sjögren's syndrome).
* Individuals with compromised immune systems, or a history of immunodeficiency disorders or undergoing immunosuppressive therapy.
* Pregnant or breastfeeding females.
* Current smokers or individuals who have quit smoking within the past 6 months.
* Individuals currently using antibiotics or have used them within the past 4 weeks.
* Individuals with a history of gastrointestinal disorders (e.g., inflammatory bowel disease, irritable bowel syndrome).
* Individuals with unstable metabolic diseases/disorders, heart failure or a history of endocarditis.
* Frequent user of alcohol or over the counter laxatives, or herbal-based supplements (but not vitamin supplements), or prescription drugs that may potentially influence the biomarkers to be measured in the study.
* Those with any chronic systemic illness that might affect participation in the trial or interpretation of results.
* Participants currently enrolled in another clinical trial involving probiotics or oral health interventions.
* Those unable to adhere to the study protocol or unlikely to complete the study period due to anticipated relocation or other personal reasons.
* Any other condition or circumstances that, in the opinion of the investigator, might compromise the safety of the participant or the validity of the study results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Effect on oral health physical condition | 3-months
  Incidence of physical abnormality in pharynx, tongue, teeth, gums and oral mucosa
Effect on other physical features | 3-months
  Incidence of any physical abnormality in the skin, eyes, ears, nose, throat, and mental health
Effect on vital signs | 3-months
  Any changes in the heart rate (heart beats per minute (bpm))
Effect on vital signs | 3-months
  Any changes in the respiratory rate (number of breaths per minute)
Effect on vital signs | 3-months
  Any changes in the blood pressure (both systolic pressure and diastolic pressure)
Effect on vital signs | 3-months
  Any changes in the body temperature
Effect on blood biochemistry | 3-months
  Any changes in the liver function tests (Serum alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase)
Effect on blood biochemistry | 3-months
  Any changes in the renal function tests (serum creatinine, serum urea, blood urea nitrogen)
Effect on blood biochemistry | 3-months
  Any changes in the lipid profile tests (serum total cholesterol, serum triglycerides, serum high density lipoprotein-cholesterol, serum low density lipoprotein-cholesterol)
Effect on blood biochemistry | 3-months
  Any changes in the blood glucose levels
Effect on blood electrolytes balance | 3-months
  Electrolyte tests (e.g., sodium, potassium, chloride, bicarbonate)
Effect on hematology | 3-months
  Full blood count
Incidence of inflammation | 3-months
  C-recative protein (CRP) blood test
Incidence of gastrointestinal side effects | 3-months
  Abdominal pain, bloating, gastric reflux, nausea, vomiting, diarrhea, and gas or flatulence
Incidence of Adverse events (AEs) | 3-months
  Any adverse events that may occur during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Jam Ghulam Qadir Civil Hospital, Hub, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Pierro F, Bugti AA, Bano A, Kara M, Ujjan I, Mumtaz N, Gull Y, Cazzaniga M, Bertuccioli A, Tanda ML, Zerbinati N, Hameed S, Khan A. Study to evaluate the safety and tolerability of Streptococcus salivarius eK12, a genetically modified strain derived from the oral probiotic S. salivarius K12: Results from a randomized, double-blind, placebo-controlled, parallel-group clinical trial. Front Nutr. 2025 Dec 8;12:1701611. doi: 10.3389/fnut.2025.1701611. eCollection 2025. PMID 41438195